CLINICAL TRIAL: NCT00354926
Title: Open-Label, Multicenter, Phase 1/2 Dose-Escalation Study of AME-133v (LY 2469298), Administered Intravenously in Four Weekly Doses, in Subjects With CD20+ Follicular Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of an Anti-CD20 Monoclonal Antibody (AME-133v) to Treat Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Molecular Evolution (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AME 06.133v.A
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; rituximab; humanized monoclonal antibody; anti-CD20 monoclonal antibody
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ocaratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AME 133v (Experimental): All subjects will receive weekly intravenous infusions of AME-133v. Each subject will receive a total of 4 infusions administered once a week for 3 consecutive weeks.
  Interventions: Biological: AME-133v (LY2469298)

INTERVENTIONS:
Biological: AME-133v (LY2469298) — IV 4X weekly X 4

SUMMARY:
This study is designed to provide evidence of the safety and a preliminary understanding of the efficacy of AME 133v.

DETAILED DESCRIPTION:
The protein engineering of AME-133v is hypothesized to result in an anti-CD20 therapy with greater potency and efficacy in all patients, but particularly in genetically defined subpopulations that respond poorly to rituximab because they express a low affinity version of the Fc receptor on their immune effector cells. A monoclonal antibody that has increased binding for this receptor should be more effective in stimulating effector cell killing and thus improve response to the antibody.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study protocol, subjects have to meet all of the following criteria.

* Have morphologically confirmed diagnosis of CD-20+ follicular B-cell non-Hodgkin's lymphoma;
* Have the low affinity form of FcγRIIIa (F/F or F/V at position 158) as determined by FcR genotyping;
* Have measurable disease. Measurable masses (such as enlarged lymph nodes) must have a clearly defined bi-dimensional diameter of at least 1.5 x 1.5 cm on physical examination or ≤ 1.5 cm in one of the dimensions by CT, MRI, or plain radiograph;
* Have received prior treatment with chemotherapy given without rituximab; OR, Have not relapsed or progressed within 120 days (inclusive) of the last infusion of rituximab;
* Be 18 years of age or greater;
* Have a negative pregnancy test, if relevant. Women of childbearing potential (not postmenopausal for at least one year and not surgically incapable of bearing children) must agree not to become pregnant for the duration of the study. To do this, they must agree to use a medically acceptable contraceptive regimen;
* Have a performance status of 0 to 2 on the ECOG performance scale;
* Have adequate hematopoietic, renal, and hepatic function defined as:

  1. Absolute neutrophil count greater than 1,500/mm³;
  2. Platelet count greater than 75,000/mm³;
  3. Hemoglobin at least 8 g/dL;
  4. Serum creatinine ≤ 1.5x upper limit of normal;
  5. Total bilirubin ≤ 1.5x upper limit of normal;
  6. ALT ≤ 1.5 x upper limit of normal;
  7. Alkaline phosphatase ≤ 1.5x upper limit of normal.
* No evidence of hepatitis B or C infection (no detectable HBV DNA or HCV RNA);
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, or other investigational therapy for at least 30 days prior to study enrollment;
* Have discontinued all high-dose corticosteroid therapy at least 30 days prior to study enrollment (≤ 10 mg/day of Prednisone or equivalent is allowable);
* Have life expectancy of more than 3 months;
* Be able to give written informed consent.

Exclusion Criteria:

Subjects with any of the following exclusions are not allowed to participate in the study.

* Allergy to monoclonal antibodies or any of the study drug components;
* Concurrent malignancy that could complicate interpretation of response evaluation, including any histologic evidence of diffuse B-cell lymphoma. Non-melanoma skin cancer and carcinoma in situ of the cervix are not exclusions;
* Significant cardiac disease (e.g. NYHA CHF of class III or IV, history of MI within one year prior to study Day 1, unstable angina, uncontrolled hypertension, clinically significant cardiac arrhythmia (CTCAE Grade 2 or higher), or clinically significant baseline ECG or MUGA abnormality.
* Positive test for serum cardiac troponins (cTnI or cTnT assay; special processing required, and the same assay must be used throughout the study; see Study Reference Manual)
* Active infection requiring oral or i.v. antibiotics;
* Administration of blood transfusions or red blood cell growth factors within 10 days preceding enrollment into the protocol;
* Administration of white cell growth factors within 28 days preceding enrollment into the protocol;
* Concomitant nonmalignant disease(s) which could interfere with implementation of the protocol, make the study results difficult to interpret, or which represent additional safety risks;
* History of HIV-associated non-Hodgkin's lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Until the patient is off study (an average of 10 months)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Link, MD, Principal Investigator — University of Iowa; Andres Forero-Torres, MD, Principal Investigator — University of Alabama Medical Center; Nam Dang, MD, Principal Investigator — Nevada Cancer Institute; Sven de Vos, MD, PhD, Principal Investigator — University of California, Los Angeles; Kristen Ganjoo, MD, Principal Investigator — Stanford University; Brad Pohlman, MD, Principal Investigator — The Cleveland Clinic; Mitchell R. Smith, MD, PhD, Principal Investigator — Fox Chase Cancer Center; Michael E. Williams, MD, Principal Investigator — University of Virginia Health Systems; Ian Flinn, MD, PhD, Principal Investigator — SCRI Development Innovations, LLC; Markus Mapara, MD, PhD, Principal Investigator — University of Pittsburgh Medical Center; Stephanie A. Gregory, MD, Principal Investigator — Rush University Medical Center
Locations (11):
- United States (11):
  - University of Alabama Medical Center, Birmingham, Alabama
  - UCLA Medical Hematology and Oncology, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Ganjoo KN, de Vos S, Pohlman BL, Flinn IW, Forero-Torres A, Enas NH, Cronier DM, Dang NH, Foon KA, Carpenter SP, Slapak CA, Link BK, Smith MR, Mapara MY, Wooldridge JE. Phase 1/2 study of ocaratuzumab, an Fc-engineered humanized anti-CD20 monoclonal antibody, in low-affinity FcgammaRIIIa patients with previously treated follicular lymphoma. Leuk Lymphoma. 2015 Jan;56(1):42-8. doi: 10.3109/10428194.2014.911859. Epub 2014 Jul 14. PMID 24717109